CLINICAL TRIAL: NCT03999320
Title: Impact of Sophrology on Exercise Capacity of Adolescents and Young Adults With Congenital Heart Disease : Multicenter Randomized Controlled Trial
Brief Title: Sophrology and Congenital Heart Disease
Acronym: SOPHRO CARE
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Montpellier (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: RECHMPL18_0043; UF7590 (Other: UH Montpellier)
Record Dates: First submitted 2019-06-24; First posted 2019-06-26 (Actual); Last update posted 2023-10-03 (Actual); Status verified 2023-10

CONDITIONS: Congenital Heart Disease
MeSH Terms: conditions — Heart Defects, Congenital

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Sophrology group (Experimental): 8 sophrology sessions, approximately 60 minutes each, spread over 12 months
  Interventions: Other: Sophrology sessions
- Control group (Other): usual care
  Interventions: Other: usual care

INTERVENTIONS:
Other: Sophrology sessions — 8 sophrology sessions, approximately 60 minutes each, spread over 12 months
  Arms: Sophrology group
Other: usual care — usual care
  Arms: Control group

SUMMARY:
The SOPHRO-CARE trial aims to measure the impact of sophrology on exercise capacity of adolescents and young adults with congenital heart disease.

Investigator hypothesized that a series of group sessions of sophrology may improve the exercise capacity, in this population.

DETAILED DESCRIPTION:
Adolescents and adults with congenital heart disease (CHD) have reduced exercise capacity compared to the general population.

Our recent randomized trial in a population of children and adolescents with asthma showed that sophrology improve lung function (NCT02114398). Sophrology, from the Greek "study of consciousness in harmony", is an adjuvant therapy, considered in healthcare as a relaxation technique, mainly based on breathing.

Investigator assume that adolescents and young adults (13-25 y.o.) with CHD who participate in a program of sophrology with structured group sessions will improve their exercise capacity as measured by the maximum oxygen uptake (VO2max), in comparison with a control group.

ELIGIBILITY:
Inclusion Criteria:

* Patient aged 13 to 25 years old
* With a congenital heart disease (CHD) as defined in the international anatomic and clinical classification (ACC) - CHD classification.
* Informed consent from adult patients or parents/legal guardians for minor patients

Exclusion Criteria:

* Medical contraindication to perform an exercise test.
* Patient already included in a clinical trial.
* Cardiac surgery planned during the study
* Severe intellectual disability that does not allow practice of sophrology exercise or questionnaires to be completed .

Ages: 13 Years to 25 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 200 (Actual)
Dates: Start 2019-07-19 (Actual); Primary Completion 2023-09-19 (Actual); Study Completion 2023-09-19 (Actual)

PRIMARY OUTCOMES:
Maximum oxygen uptake (VO2 max) | Variation between Baseline (M0) and at 12 months (M12)
  VO2max Variation

SECONDARY OUTCOMES:
Quality of life score | Evolution of the PedsQL 4.0 self-reported scores from month 0 to month 12
  Quality of life score variation (PedsQL, 24 items), range score from 0 to 100, higher score indicating better quality of life.
Physical activity score | Variation between Baseline (M0) and at 12 months (M12)
  Score of physical activity (Ricci and Gagnon questionnaire, 9 items, total range score from 6 to 45, higher score indicating a higher level of physical activity)

CONTACTS AND LOCATIONS:
Overall Officials: Pascal AMEDRO, MD, Principal Investigator — UH Montpellier; Sophie GUILLAUMONT, MD, Principal Investigator — Saint Pierre Institut; Yves DULAC, MD, Principal Investigator — UH Toulouse; Damien BONNET, MD, Principal Investigator — APHP Necker; Alban Louen BARUTEAU, Professor, Principal Investigator — UH Nantes
Locations (2):
- France (2):
  - CHU de Montpellier, Montpellier, Occitanie
  - Institut Saint-Pierre, Palavas-les-Flots

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Moreau J, Lavastre K, Romieu H, Charbonnier F, Guillaumont S, Bredy C, Abassi H, Werner O, De La Villeon G, Requirand A, Auer A, Matecki S, Karsenty C, Guitarte A, Hadeed K, Dulac Y, Souletie N, Acar P, Bajolle F, Bonnet D, Negre-Pages L, Mura T, Mounier M, Seguela PE, Thomas J, Iriart X, Jean-Benoit-Thambo, Amedro P. Impact of Sophrology on cardiopulmonary fitness in teenagers and young adults with a congenital heart disease: The SOPHROCARE study rationale, design and methods. Int J Cardiol Heart Vasc. 2020 Mar 3;27:100489. doi: 10.1016/j.ijcha.2020.100489. eCollection 2020 Apr. PMID 32154361
- See also: Impact of Sophrology on cardiopulmonary fitness in teenagers and — http://creativecommons.org/licenses/by/4.0/